CLINICAL TRIAL: NCT06418698
Title: The Prediction of Intracranial Artery Calcification on Adverse Outcomes of Large Vessel Occlusive, Acute Ischemic Stroke Patients After Mechanical Thrombectomy: A Prospective Cohort, Observational Study
Brief Title: The Correlation of Intracranial Artery Calcification and Outcomes of Mechanical Thrombectomy
Acronym: CAIS-MT
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LC2024ZD026
Record Dates: First submitted 2024-04-06; First posted 2024-05-17 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Stroke, Acute; Ischemic Stroke; Vascular Diseases; Central Nervous System Diseases; Nervous System Diseases; Stroke; Brain Diseases; Cerebrovascular Disorders; Intracranial Arterial Calcification
Keywords: Acute ischemic stroke; Large vessel occlusion; Mechanical thrombectomy; Endovascular treatment; Agatston score; Prospective cohort study; Intracranial atherosclerotic disease
MeSH Terms: conditions — Stroke; Ischemic Stroke; Vascular Diseases; Central Nervous System Diseases; Nervous System Diseases; Brain Diseases; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with acute ischemic stroke due to large or medium vessel occlusion: Patients with acute ischemic stroke due to large or medium vessel occlusion meeting inclusion criteria, must accept mechanical thrombectomy and have CT images which can get the IAC Agatston score.

SUMMARY:
CAIS-MT is a single-center, prospective cohort study, to evaluate the correlation between outcomes of endovascular treatment(EVT) and intracranial artery calcification(IAC) in patients with acute ischemic stroke due to large or medium vessel occlusion.

DETAILED DESCRIPTION:
This study have to objective to evaluate the predictive value of IAC Agatston score in patients with acute ischemic stroke due to large or medium vessel occlusion on worse angiographic and functional outcomes after EVT. The result of this study will provide a upfront basis for risk stratification of adverse outcomes of EVT by using quantitative IAC, so as to get a reference for an individualized and precise plan of EVT.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant women with acute stroke symptoms aged over 18 years.
* Occlusion of the intracranial internal carotid artery, the middle cerebral artery, the anterior cerebral artery, the posterior cerebral artery, basilar artery and intracranial vertebral artery confirmed by CT, MR angiography, or digital subtraction angiography.
* No absolute contraindication to iodinated contrast media.
* Planned treatment with EVT by clinical care team.
* Informed consent obtained from patients or their legal representatives.
* Willing to be followed up as required by the clinical study protocol.

Exclusion Criteria:

* Acute ischemic stroke occurs over 24 hours of time last known well.
* Neurologic deficits caused by diagnoses other than ischemic stroke, such as intracerebral hemorrhage, subarachnoid hemorrhage, or intracranial tumors.
* With other underlying factors leading to IAC, such as hyperthyroidism, end-stage renal disease, long-term oral intake of vitamin K antagonist(Warfarin), chronic vitamin D deficiency or overdose, persistent hypomagnesemia, persistent hypercalcemia, persistent hyperphosphatemia and high oral calcium intake.
* Lack of non-contract CT images on admission and significant artifacts in CT images preventing IAC measurement.
* Severe renal insufficiency (estimated glomerular filtration rate < 30ml/min or serum creatinine > 220μmol/L (2.5mg/dl)).
* Previous cerebrovascular intervention treatment or craniotomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of acute ischemic stroke due to large or medium vessel occlusion, who are enrolled at Zhujiang Hospital and meet the indication for EVT.
Sampling Method: Non-Probability Sample
Enrollment: 434 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a adverse functional outcome at 3 months | 90(±7) days
  Modified Rankin Scale(mRS) score > 2

SECONDARY OUTCOMES:
Proportion of patients without disability at 3 months | 90(±7) days
  mRS score 0-1
Proportion of patients with functional independence at 3 months | 90(±7) days
  mRS score 0-2
Proportion of patients ambulatory or bodily needs-capable or better at 3 months | 90(±7) days
  mRS score 0-3
Change of the NIHSS score at 24 hours from baseline | 24 hours
  Change of the NIHSS score at 24 hours from baseline
Change of the NIHSS score at 6 days or discharge if earlier from baseline | 6(±1) days
  Change of the NIHSS score at 6 days or discharge if earlier from baseline
Health-related quality of life at 3 months | 90(±7) days
  Health-related quality of life is assessed with the European Quality Five Dimensions Five Level scale (EQ-5D-5L)
Proportion of substantial reperfusion at final angiogram | 0 day
  Substantial reperfusion is defined as a expanded Treatment in Cerebral Infarction score of 2b50 (50 to 67% reperfusion), 2b67 (67 to 89% reperfusion), 2c(90 to 99% reperfusion) or 3 (complete reperfusion)
Proportion of substantial reperfusion at final angiogram without any rescue methods | 0 day
  Substantial reperfusion is defined as a expanded Treatment in Cerebral Infarction score of 2b50 (50 to 67% reperfusion), 2b67 (67 to 89% reperfusion), 2c(90 to 99% reperfusion) or 3 (complete reperfusion)
Proportion of substantial reperfusion at first angiogram | 0 day
  Substantial reperfusion is defined as a expanded Treatment in Cerebral Infarction score of 2b50 (50 to 67% reperfusion), 2b67 (67 to 89% reperfusion), 2c(90 to 99% reperfusion) or 3 (complete reperfusion)
Proportion of patients with Symptomatic intracranial hemorrhage(sICH) within 48 hours | Within 48 hours
  ICH will be evaluated according to the Heidelberg Bleeding Classification. sICH is diagnosed if the new observed ICH is associated with any of the following conditions: 1) NIHSS score increased more than 4 points than that immediately before worsening; 2) NIHSS score increased more than 2 points in one category; 3) Deterioration led to intubation, hemicraniectomy, external ventricular drain placement or any other major interventions. Additionally, the symptom deteriorations could not be explained by causes other than the observed ICH.
Proportion of patients with any ICH within 48 hours | Within 48 hours
  ICH will be evaluated according to the Heidelberg Bleeding Classification.
Mortality at 3 months | 90(±7) days
  Mortality rates are defined as the number of deaths observed divided by the number of subjects observed over the 90-day study period.
Incidence of serious adverse events | Within 3 years
  Including but not limited to acute respiratory failure, severe or malignant cerebral artery infarction, acute heart failure, debridement decompression, and other major medical events that can result in death, immediately life-threatening, hospitalization or prolongation of this hospitalization, terminally or severely disabling/incapacitating, the loss of a significant ability to maintain normal life functioning, or medical intervention to avoid the above outcomes.
Procedure-related complications | Up to 24 hours
  such as arterial perforation, iatrogenic arterial dissection, embolization in previously uninvolved vascular territory, arterial access site hematoma, and retroperitoneal hematoma. Arterial perforation will be defined at angiography by the operator and associated with subarachnoid hemorrhage. Iatrogenic arterial dissection will be defined at angiography by the operator. Arterial access site hematoma will be assessed as a complication of arterial access puncture and defined by clinical examination and anatomic imaging. Retroperitoneal hematoma will be assessed as a complication of groin puncture and defined by imaging (ultrasound or CT or MR angiography). The definition of embolization in previously uninvolved vascular territory is noted after recanalization of the primary occlusion site, any vessel occlusions distal from the primary occlusion site are considered emboli due to periprocedural thrombus fragmentation.
Proportion of patients with new cerebrovascular events related with previous vessel occlusion at 1 year | 365(±30) days
  New cerebrovascular events are defined as progression of ischemic lesion or newly hemorrhagic lesion.
Proportion of patients with new cerebrovascular events related with previous vessel occlusion at 3 years | 1095(±30) days
  New cerebrovascular events are defined as progression of ischemic lesion or newly hemorrhagic lesion.
Proportion of patients with new cerebrovascular events irrelated with previous vessel occlusion at 1 year | 365(±30) days
  New cerebrovascular events are defined as progression of ischemic lesion or newly hemorrhagic lesion.
Proportion of patients with new cerebrovascular events irrelated with previous vessel occlusion at 3 years | 1095(±30) days
  New cerebrovascular events are defined as progression of ischemic lesion or newly hemorrhagic lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Duan Chuanzhi, MD, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No